CLINICAL TRIAL: NCT01433861
Title: Phase III Prospective Randomized Clinical Trial of Laparoscopy-assisted Proximal Gastrectomy (LAPG) and Laparoscopy-assisted Total Gastrectomy (LATG) for Upper Gastric Cancer. (Multicenter Study)
Brief Title: Laparoscopy-assisted Proximal Gastrectomy Versus and Laparoscopy-assisted Total Gastrectomy
Acronym: PRAPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: We planed to study later
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBHGS
Record Dates: First submitted 2011-09-10; First posted 2011-09-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; proximal gastrectomy; total gastrectomy; laparoscopy; reflux esophagitis; double tract reconstruction
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAPG (Active Comparator): LAPG : laparoscopy-assisted proximal gastrectomy with double tract reconstruction group
  Interventions: Procedure: Laparoscopy-assisted gastrectomy
- LATG (Active Comparator): LATG : laparoscopy-assisted total gastrectomy group
  Interventions: Procedure: Laparoscopy-assisted gastrectomy

INTERVENTIONS:
Procedure: Laparoscopy-assisted gastrectomy — Laparoscopy-assisted proximal gastrectomy versus Laparoscopy-assisted total gastrectomy

SUMMARY:
The choice of surgical strategy for patients with proximal gastric cancer is controversial mainly because proximal gastrectomy is infamous for high rates of reflux symptoms and anastomotic stricture. but there are no prospective randomized trials until now.

The primary end point of this study is whether the rate of reflux esophagitis is different or not between LAPG and LATG. Through this study, we

DETAILED DESCRIPTION:
Prospective Randomized Clinical Trials between Laparoscopy-assisted Proximal Gastrectomy and Laparoscopy-assisted Total Gastrectomy.

LAPG reconstruction: double tract reconstruction (3 anastomosis, intracorporeal Roux-en Y esophago-jejunostomy, extracorporeal gastro-jejunostomy 10cm below esophago-jejunostomy,extracorporeal jejuno-jejunostomy 20cm below gastro-jejunostomy)

LATG reconstruction: intracorporeal Roux-en Y esophago-jejunostomy

Primary end point : incidence of reflux esophagitis after operation

Sample Size : LAPG 97 cases, LATG 97 cases (p1=0.018 p2=0.018, a=0.05, b=0.80) Non-inferiority test, non-inferior margin (delta) : 0.05. Sample size calculated by our MRCC(Medical Research Collaborating Center, http://mrcc.snubh.org)

Study duration : 48 months (enrollment 36months, follow-up 12months)

Reflux esophagitis evaluation methods

1. Ambulatory 24hr-pH esophageal holter monitoring for acid reflux
2. DISIDA scan for bile reflux
3. Endoscopic evaluation (Grading according to LA classification)
4. Visick score (subjective symptoms)
5. EORTC sto 22 and GIQLI evaluation (Quality of Life)
6. Nutritional Benefits (Body weight, Triceps Skin folds Thickness, Blood test)
7. Upper gastrointestinal study
8. Gastric emptying scan

ELIGIBILITY:
Inclusion Criteria:

* Age 20~80
* Informed consent
* No other malignancies
* Proximal gastric cancer met by following conditions

  1. Lesion located on proximal stomach (upper one third)
  2. Lesion below 5cm in size
  3. Lesion confined to proper muscle depth (cT2)
  4. No evidence of metastatic enlarged LN on #5, 6, 4d, 10 basins and other distant metastasis. (cN1)

Exclusion Criteria:

* If patients is only suitable to total gastrectomy, he will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of reflux esophagitis | postoperative 3 month
  Comprehesive evaulation by 24hr pH monitoring, DISIDA scan, Endoscopic evaluation according to LA classification and Visick score
Rate of reflux esophagitis | postoperative 6 month
  Comprehesive evaulation by 24hr pH monitoring, DISIDA scan, Endoscopic evaluation according to LA classification and Visick score
Rate of reflux esophagitis | postoperative 12 month
  Comprehesive evaulation by 24hr pH monitoring, DISIDA scan, Endoscopic evaluation according to LA classification and Visick score

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Ho Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyenggi, South Korea

IPD SHARING:
Plan to Share IPD: No